CLINICAL TRIAL: NCT01070459
Title: The Effect of an Aerobic Training Programme on the Aerobic Capacity, Functional Behavior and the Cardiovascular Risk Factors in Stroke Patients
Brief Title: The Effect of an Aerobic Exercise Programme in Stroke Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University College of Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); KU Leuven (Other); University Hospital, Antwerp (Other)
Responsible Party: University College of Antwerp, Campus HIKE Merksem
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B30020107752
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke aerobic exercise daily functioning rehabilitation
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control group (Placebo Comparator): The patients continue their regular therapy in the rehabilitation center. They participate in a 12-week programme of passive mobilisation of the hemiplegic knee, using a continuous passive motion device. Patients will be trained three times a week, 30 minutes/session.
  Interventions: Behavioral: Follow-up control group
- Aerobic exercise group (Experimental): The patients continues their regular therapy in the rehabilitation center. They participate in a 12-week programme of aerobic training 30 minutes/session, using a leg cycle bike. Patients will be trained three times a week. The heart rate will vary from 50 tot 75% of their predicted heart rate. Each patient will be provided with an progressive exercise prescription based on 50-75% of their predicted maximum heartrate. Throughout the training sessions the heart rate will be monitored continuously with a polar pulse rate. Within these 12 week training programme 4 information sessions will be offered to patients and relatives about risk factors of stroke, usefulness of an active lifestyle and healthy eating.
  Interventions: Behavioral: Aerobic exercise group; Behavioral: Follow-up first aerobic exercise group; Behavioral: Follow-up second aerobic exercise group
- Follow-up first aerobic exercise group (Experimental)
  Interventions: Behavioral: Follow-up first aerobic exercise group
- Follow-up control group (Placebo Comparator)
  Interventions: Behavioral: Control group; Behavioral: Follow-up control group
- Follow-up second aerobic exercise group (Experimental)
  Interventions: Behavioral: Follow-up second aerobic exercise group

INTERVENTIONS:
Behavioral: Aerobic exercise group — The patients continue their regular therapy in the rehabilitation center. They participate in a 12-week programme of aerobic training 30 minutes/session, using a leg cycle bike. Patients will be trained three times a week. The heartrate will vary from 50 tot 75% of their predicted heart rate. Each patient will be provided with an progressive exercise prescription based on 50-75% of their predicted maximum heartrate. Throughout the training sessions the heart rate will be monitored continuously with a polar pulse rate. Within these 12 week exercise programme four information sessions will be offered to patients and relatives about risk factors of stroke, usefulness of an active lifestyle and healthy eating.
  Arms: Aerobic exercise group
Behavioral: Control group — The patients continue their regular therapy in the rehabilitation center. They participate in a 12-week programme of passive mobilisation of the hemiplegic knee, using a continuous passive motion device. Patients will be trained three times a week, 30 minutes/session.
  Arms: Follow-up control group
Behavioral: Follow-up first aerobic exercise group — The experimental aerobic exercise will be divided in two groups at random after the 12 weeks aerobic exercise programme. The first group will get feedback on how to train further their aerobic capacity within the following 9 months. The second group will not undergo the feedback programme.
  Arms: Aerobic exercise group; Follow-up first aerobic exercise group
Behavioral: Follow-up control group — No intervention will be offered in a period of 9 months after the passive mobilisation programme
  Arms: Control group; Follow-up control group
Behavioral: Follow-up second aerobic exercise group — The experimental aerobic exercise will be divided in two groups at random after the 12 weeks aerobic exercise programme. The second group will not undergo the feedback programme. This group will be measured but not treated with an intervention programme
  Arms: Aerobic exercise group; Follow-up second aerobic exercise group

SUMMARY:
This study aims to investigate the effect of aerobic exercise on the aerobic capacity, the daily functioning, post-stroke fatigue , depression and cardiovascular risk factors in stroke patients.

DETAILED DESCRIPTION:
People with neurologic impairments after stroke often show decreased aerobic exercise capacity. The etiologies of which are assigned to physiologic changes in paretic muscle, gait deficits and disability-related deconditioning. This declares that stroke patients live an inactive lifestyle and therefore stay cardiovascular risk patients.

The usefulness of aerobic training on aerobic capacity is recently been proved in clinical stroke research. However, no study can shown the long-term effect of aerobic exercises. Also the effect of aerobic exercises on daily functioning, fatigue and depression in stroke needs to be established.

ELIGIBILITY:
Inclusion Criteria:

* First CVA according to the WHO definition (A primary, first ever stroke ash revealed by rapidly developing clinical signs or focal or global disturbance or cerebral function, with symptoms lasting 24 hours or longer or leading to death, with no apparent cause other than or vascular origin.) This includes ischemic infarct or an intracerebral haemorrhage
* The offense can be maximum 3 up to 6 weeks after onset
* Patient must be able to follow simple verbal instructions
* To cycle during 1 minute at 20 Watt, 50RPM,
* Cardiac stable

Exclusion Criteria:

* Have another neurological impairments with permanent damage such as former cranial trauma, multiple sclerosis, epileptic status… which already present were for current CVA
* Having on CVA resembling symptoms as a result of subdural haemorrhage, a tumour, encephalitis or a trauma
* Barthel index < 50 before the stroke onset
* Age > 80 year
* No authorisation form of the patient or of the family
* Absolute contra-indications for effort test (ACC/AHA guidelines)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
VO2-peak, strength, walking, activities of daily living | baseline , after 12 weeks training. Follow-up measurements after 6 months, 1 and 2 years after baseline.

SECONDARY OUTCOMES:
post-stroke fatigue, depression, lifestyle, cardiovascular risk factors | baseline , after 12 weeks training. Follow-up measurements after 6 months, 1 and 2 years after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cras, prof. dr., Study Chair — Universiteit Antwerpen; Yves Vanlandewijck, prof.dr., Study Director — KU Leuven; Hilde Feys, prof.dr., Study Director — Catholic University of Antwerp; Steven Truijen, dr., Study Director — University college Antwerp; Dirk Vissers, dr., Study Director — University College of Antwerp; christel Vanroy, PhD, Principal Investigator — University College Antwerp
Locations (1):
- Revalidatiecentrum Sint-Ursula, Herk-de-Stad, Limburg, Belgium

REFERENCES:
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Vanroy C, Vanlandewijck Y, Cras P, Truijen S, Vissers D, Swinnen A, Bosmans M, Wouters K, Feys H. Does a cycling program combined with education and followed by coaching promote physical activity in subacute stroke patients? A randomized controlled trial. Disabil Rehabil. 2019 Feb;41(4):413-421. doi: 10.1080/09638288.2017.1395084. Epub 2017 Nov 5. PMID 29105516
- [Derived] Vanroy C, Feys H, Swinnen A, Vanlandewijck Y, Truijen S, Vissers D, Michielsen M, Wouters K, Cras P. Effectiveness of Active Cycling in Subacute Stroke Rehabilitation: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1576-1585.e5. doi: 10.1016/j.apmr.2017.02.004. Epub 2017 Mar 8. PMID 28284834